CLINICAL TRIAL: NCT02514954
Title: Postprandial Blood Glucose Control With BioChaperone® Combo and Insulin Lispro (Humalog®) Mix 25 in People With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BC3-CT019
Record Dates: First submitted 2015-07-29; First posted 2015-08-04 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BioChaperone® Combo (Experimental): 1 single dose 400 U/mL
  Interventions: Drug: Biochaperone® Combo
- Humalog® Mix25 (Active Comparator): 1 single dose 100 U/mL
  Interventions: Drug: Humalog® Mix25

INTERVENTIONS:
Drug: Biochaperone® Combo — Subcutaneous injection of an individualized dose
  Arms: BioChaperone® Combo
Drug: Humalog® Mix25 — Subcutaneous injection of an individualized dose
  Arms: Humalog® Mix25

SUMMARY:
Each subject will be randomly allocated to a sequence of two treatments applied at two separate dosing visits. At each dosing visit subjects will be injected with individualised doses of either BioChaperone® Combo or Humalog® Mix 25 immediately before ingesting a standardised mixed meal [(t=0 min) start of the meal]. Insulin doses will be identical at both dosing visits of one individual and will be administered subcutaneously in the abdominal region. Subjects will be asked to consume a standardised meal (e.g. pizza) for dinner at home in the evening before each dosing visit. Subjects will attend the clinical site in a fasted state in the morning of each dosing day and stay at the clinical trial centre until 10-hour after dosing (standardised test-meal procedure has been terminated after 6h). The two dosing visits will be separated by a wash-out period of 5-15 days.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) >= 12 months.
* Treated with multiple daily insulin injections or CSII >= 12 months.
* Current total daily insulin treatment < 1.2 (I)U/kg/day.
* Current total daily bolus insulin treatment < 0.7 (I)U/kg/day.
* Usual Insulin bolus dose between 0.8 and 2 (I)U per 10 g CH (both inclusive). Expecting prandial insulin dose range for standardised meal test between 5 and 12 (I)U.
* BMI 18.5-28.0 kg/m^2 (both inclusive).
* HbA1c <= 9.0% by local laboratory analysis
* Fasting C-peptide <= 0.3 nmol/L.

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products.
* Type 2 diabetes mellitus.
* Previous participation in this trial. Participation is defined as randomised.
* Participation in any Clinical Trial within 3 months prior to this trial.
* Clinically significant abnormal haematology, biochemistry, lipids, or urinalysis screening tests, as judged by the Investigator considering the underlying disease.
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea), as judged by the Investigator.
* Known slowing of gastric emptying and or gastrointestinal surgery that in the opinion of the investigator might change gastrointestinal motility and food absorption.
* Unusual meal habits and special diet requirements or unwillingness to eat the food provided in the trial.
* Women of child bearing potential, not willing to use contraceptive methods.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Delta AUCBG,0-2h | 2 hours
  Incremental area under the blood glucose concentration-time curve from 0-2 hours after a standardised meal

SECONDARY OUTCOMES:
Delta AUCBG,0-6h | 6 hours
  Incremental area under the blood glucose concentration-time curve from 0-6 hours after a standardised meal
BGmax | 6 hours
  Maximum blood glucose concentration after a standardised meal (0-6 hours)
tBGmax | 6 hours
  Time to maximum blood glucose concentration after a standardised meal (0-6 hours)
AUCLisp,0-6h, | 6 hours
  Area under the plasma insulin lispro concentration-time curve from 0-6 hours
AUCGlarg,0-6h | 6 hours
  Area under the plasma insulin glargine concentration-time curve from 0-6 hours
Cmax,Lisp | 6 hours
  Maximum observed plasma insulin lispro concentration
Cmax,Glarg | 6 hours
  Maximum observed plasma insulin glargine concentration
Adverse events | Up to 7 weeks
  Number of adverse events
Local tolerability | Up to 7 weeks
  Number and intensity of injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, MD, Principal Investigator — Profil Institut Für Stoffwechselfforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany